CLINICAL TRIAL: NCT05060770
Title: Transcriptiomic Analysis of Inflammatory Bowel Disease-associated Colorectal Cancer. A French Retrospective Study of 26 Cases Identified at the Nancy University Hospital
Brief Title: Transcriptomic Study of IBD-associated Colorectal Cancer
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, MULLER Marie, Doctor (MD, PhD Student), Principal investigator, Central Hospital, Nancy, France
Other Study IDs: 2021PI125
Record Dates: First submitted 2021-09-19; First posted 2021-09-29 (Actual); Last update posted 2021-10-07 (Actual); Status verified 2021-09

CONDITIONS: Colorectal Cancer, Genetics of
Keywords: inflammatory bowel disease
MeSH Terms: conditions — Colorectal Neoplasms; Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Genetic: transcriptomic analysis — transcriptomic analysis on preserved tumor tissue

SUMMARY:
Chronic inflammatory bowel disease (IBD) is associated with an increased risk of colorectal cancer (CRC) in historical cohorts. The pathways of oncogenesis of these CRCs, which are very different clinically from de novo CRCs, are currently unknown. The aim of our work is to identify specific molecular signatures of CRC occurring in the setting of IBD.

ELIGIBILITY:
Inclusion Criteria:

* Person 18 years of age or older
* Person with colorectal cancer in the context of IBD
* Person who has received complete information on the organization of the research and who has signed an informed consent
* Person affiliated to a social security plan or beneficiary of such a plan.

Exclusion Criteria:

* Person referred to in articles L. 1121-5, L. 1121-7 and L1121-8 of the public health code:
* Pregnant woman, parturient or nursing mother
* Minor (not emancipated)
* Adult person subject to a legal protection measure (guardianship, curatorship, safeguard of justice)
* Person of legal age who is unable to express his or her consent
* Person deprived of liberty by a judicial or administrative decision, persons subject to psychiatric care under articles L. 3212-1 and L. 3213-1.

Ages: 18 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: >/= 18 years old patient operated on at the Nancy university hospital for IBD associated CRC
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2010-01-01 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
IBD associated CRC oncogenesis | 1 year
  Percentage of gene expression variation in CRC tumor tissue samples in the following groups patients with CRC and IBD

IPD SHARING:
Plan to Share IPD: No